CLINICAL TRIAL: NCT01211119
Title: Novel One-step Repair of Knee Meniscal Tear Using Platelet-rich Fibrin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Wing P. Chan, Wan Fang Hospital Department of Radiology
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99022
Record Dates: First submitted 2010-09-20; First posted 2010-09-29 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Meniscal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- platelet-rich fibrin, PRF (Experimental)
  Interventions: Other: No PRF

INTERVENTIONS:
Other: No PRF — Group B (n=6), implantation of PRF after partial menisectomy and suture; Group (n=6), partial menisectomy only

SUMMARY:
Currently, most knee meniscal tears are treated by partial or complete meniscectomy, or by suture repair when it is possible. Recently, the investigators have successfully developed and implanted a novel biomaterial, platelet-rich fibrin (PRF), to treat articular cartilage defect in pigs. The PRF is autogenesis as a natural fibrin-based biomaterial favorable to the development of microvascularization and enables local and progressive delivery of growth factors providing unique properties for tissue remodeling and wound healing. The advantages of using PRF implantation include no transplant rejection and no need to perform second operation. Knee meniscal repair using PRF has not been reported before. The aim of this study is to investigate whether PRF implantation can facilitate regeneration process of meniscectomized knee and T2-map MRI can monitor the process in those patients with meniscal tears.

A total of 18 adult patients with torn menisci (outer 1/3, posterior horn, medial meniscus) will be recruited and randomly divided into three groups: A (n=6), implantation of PRF after partial menisectomy; B (n=6), implantation of PRF after partial menisectomy and suture; C (n=6), partial menisectomy only. All studied knee will be scanned on a 1.5-T MRI with surface coil at baseline before surgery, 3 months and 6 months and 12 months after surgery.

The investigators believe that PRF enables to facilitate regeneration of meniscectomized knee, and T2-map MRI enables monitoring healing process of meniscal tears.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 45 years old;
* time of injury to surgery within 8 weeks
* patients who will sign inform consent
* patients with clinical and MRI diagnosis of meniscal tears who will undergo arthroscopy
* patients who will make MRI diagnosis at 3, 6, 12 months

Exclusion Criteria:

* major trauma
* coexist ligamentous rupture
* knee dislocations

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
MRI T2-map values in healing menisci | one-month

CONTACTS AND LOCATIONS:
Overall Officials: Wing P. Chan, Principal Investigator — Taipei Medical University-Wan Fang Hospital
Locations (1):
- Taipei Medical University-Wan Fang Hospital, Taipei, Taiwan